CLINICAL TRIAL: NCT05783115
Title: Multicentre Study on Diabetic Foot Treatment by Tibial Transportation Combined With Autologous Mesenchymal Stem Cells Local Infusion
Brief Title: Multicentre Study on Diabetic Foot Treatment
Acronym: MSDFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Second Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HANQINGLIN
Record Dates: First submitted 2023-03-06; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot; Tibial Transportation; Autologous mesenchymal stem cells Local Infusion
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibial Transportation (Active Comparator): Tibial Transportation
  Interventions: Procedure: Tibial Transportation
- Tibial Transportation Combined With Autologous mesenchymal stem cells Local Infusion (Experimental): Tibial Transportation Combined With Autologous mesenchymal stem cells Local Infusion
  Interventions: Procedure: Tibial Transportation Combined With Autologous mesenchymal stem cells Local Infusion

INTERVENTIONS:
Procedure: Tibial Transportation Combined With Autologous mesenchymal stem cells Local Infusion — transverse bone transport with bone marrow cell transplantation
  Arms: Tibial Transportation Combined With Autologous mesenchymal stem cells Local Infusion
Procedure: Tibial Transportation — transverse bone transport
  Arms: Tibial Transportation

SUMMARY:
With a rapidly growing incidence rate and a high disability rate,The Diabetic Foot has long been difficult to treatment, which has caused a huge burden to patients and society. The blood supply disorder is one of the main reasons that lead to the morbidity and difficulty in healing of diabetes feet, but there is still a lack of particularly effective treatment to improve the blood supply of diabetes feet. Both transverse bone transport and bone marrow cell transplantation have shown some clinical effects. However, the difference in efficacy between the two has not been reported. In this study, investigators compared the therapeutic effects of these two methods on the healing of diabetes foot ulcers through a controlled clinical study.

DETAILED DESCRIPTION:
In this study, investigators compared the therapeutic effects of Tibial Transportation Combined With Autologous mesenchymal stem cells Local Infusion on the healing of diabetes foot ulcers through a controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms: Wagner stage 2 or above foot ulcer (deep ulcer, abscess or osteomyelitis; localized gangrene, characterized by ischemic gangrene, usually with neuropathy; gangrene of the whole foot), may be accompanied by chronic limb pain, intermittent claudication, cold sensation, abnormal skin sensation and other symptoms
* Have not taken reserpine in the past week or can change to other antihypertensive drugs
* Voluntary participation and signing of informed consent

Exclusion Criteria:

* Patients with organ failure diagnosed by doctors in the past: such as heart failure, liver and kidney failure
* Patients with myocardial infarction diagnosed by doctors in the past
* With congenital or acquired organic heart disease
* With basic disease is in the active stage, such as newly diagnosed leukemia patients, or leukemia patients with relapse and refractory
* Active infection: pulmonary infection, intestinal infection and other existing infections
* Severe anemia
* Severe osteoporosis
* Have undergone amputation of both lower limbs
* The investigator judged that it was not suitable to participate in this study, including the existence of abnormal laboratory test results or clinical abnormal symptoms/signs
* There are any of the following conditions that may limit the patient's compliance or hinder data collection: dementia; Serious mental disorder, unable to express will; Unable to complete the research evaluation as required
* Other contraindications of anesthesia or surgery

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 3 months after surgery
  Visual analog scale (VAS) and its corresponding visual analog pain scale, is a psychometric scale that is generally used in hospitals and clinics by doctors to conduct pain scale surveys to understand varying degrees of pain or discomfort experienced by a patient.VAS ranges from 0 to 10 and a higher score means worse outcome.

SECONDARY OUTCOMES:
ulcer area | 3 months after surgery
  ulcer area will be record in cm2. Use a digital camera to photograph each chronic skin ulcer wound at a fixed height and angle, and use a ruler as a marker. Each photo was measured 3 times using NIH ImageJ software and analyzed using a ruler as a scale. Import the pictures collected by the digital camera into the computer, select the clearest picture, apply the NIH ImageJ software, use a tracer pen to sketch the contour of the ulcer surface along the edge of the ulcer, and obtain the pixel square value. At the same time, use a tracer pen to sketch the linear distance of 1 cm on the scale, to obtain the pixel value of 1 cm linear distance, and then multiply the pixel value of 1 cm to obtain. The pixel square value of 1 cm2 is divided by the pixel square value of the ulcer surface contour to obtain the chronic ulcer skin area.
Wagner grade | 3 months after surgery
  The Wagner Diabetic Foot Ulcer Grade Classification System. The Wagner diabetic foot ulcer classification system assesses ulcer depth and the presence of osteomyelitis or gangrene by using the following grades.Wagner grade ranges from 0 to 10 and a higher score means worse outcome.
Painless walking distance | 3 months after surgery
  Painless walking distance
Ankle brachial index | 3 months after surgery
  a simple test that compares the blood pressure in the upper and lower limbs
skin temperature | day after surgery
  skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Qinglin Han, Dr, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of nantong university, Nantong, Jiangsu, China